CLINICAL TRIAL: NCT01235780
Title: Factors Affecting Corneal Hysteresis in Taiwanese
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shih-Hong Huang MD,PhD, Research Ethics Review Committee of Far Eastern Memorial Hospital
Other Study IDs: 098060-3
Record Dates: First submitted 2010-08-08; First posted 2010-11-08 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2009-12

CONDITIONS: Corneal Hysteresis
Keywords: corneal hysteresis, ocular response analyzer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate the factors affecting corneal hysteresis (CH) in Taiwanese.

DETAILED DESCRIPTION:
The ocular response analyzer (ORA, Reichert Ophthalmic Instruments, Buffalo, NY, USA) measures the biomechanical properties of the cornea in vivo. It provides several measurements including CH, corneal resistance factor (CRF), corneal-compensated intraocular pressure (IOPcc), and Goldmann-correlated intraocular pressure (IOPg). Corneal hysteresis is described as the viscous damping due to the viscoelastic resistance of the cornea to a deformation pulse by an air jet of the tonometer. Whereas CH may reflect corneal viscosity, the CRF may relate to the elastic properties of the cornea. Both parameters are measured by the ORA using a dynamic bidirectional process.

CH can be affected by various ocular disorders and operation. In previous studies, CH was found to be significantly lower in keratoconus, Fuchs' dystrophy, and glaucoma. After laser in situ keratomileusis (LASIK) and phacoemulsification, CH permanently or temporally decreased. Among normal population, CH was also variable and associated with several factors: age, gender, intraocular pressure, central corneal thickness, and corneal curvature. High myopic patients with long axial length were found to have lower CH than in normal subjects. CH can also affected by races, and CH was largely discussed in Caucasian population. Herein we studied normal population of CH and associated factors and in Taiwan.

We are planned to conduct a retrospective study from January to July, 2009 at Department of Ophthalmology, Far Eastern Memorial Hospital, Taipei, Taiwan by chart review. We will enroll the patients with bilateral cataract, or unilateral cataract and healthy fellow eye, who not having other ocular pathology, prior ocular surgery, or previous trauma. Several ocular parameters and demographics of both un-operated eyes in these patients are measured. CRF, IOPcc, IOPg, and CH are measured by ORA. Central corneal thickness is measured using the ORA's integrated handheld ultrasonic pachymeter. The IOLMaster (Carl Zeiss, Jena, German) is used to obtain the ocular biometry including axial length, anterior chamber depth, and keratometry. Linear regression models were used to test the correlation of CH and quantitative factors. The chi-square test was used to find the significance of correlation in categorical values.

One or two eyes of the patients undergoes uneventful phacoemulsification and in-the-bag implantation of posterior chamber intraocular lens (one-piece AcrySof, Alcon lab, Texas, USA) by one surgeon (Wang JK). The sutureless corneal wound was 2.75 mm long. CRF, IOPcc, IOPg, and CH are measured by ORA preoperatively and 1 day, 1 week, 2 weeks, 3 weeks, 1 month, 2 months, and 3 months postoperatively. Paired t test was used to compare the changes of these parameters following the operation.

We expect that some factors will correlate with CH, such as axial length, IOP, age, and central corneal thickness. Temporary reduction in CH is possibly shortly after phacoemulsification, and returning to the baseline following a period of time.

ELIGIBILITY:
Inclusion Criteria:

* normal population

Exclusion Criteria:

* no other ocular diseases except cataract, no prior ocular operation, no prior ocular trauma

Ages: 33 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal population and patients receiving phacoemulsification
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2009-12; Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kang Wang, M.D., Study Chair — Ophthalmologic Department, Far Eastern Memorial Hospital